CLINICAL TRIAL: NCT06941324
Title: SFBT for AYA Cancer Survivors' Psychological Distress: Evaluating Solution-Focused Brief Therapy as a Strength-Based Psychotherapeutic Intervention for Psychological Distress in Adolescents and Young Adults With Cancer
Brief Title: Solution-Focused Brief Therapy for Support of Psychological Distress in Adolescent and Young Adult Cancer Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Children's Cancer Research Fund (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UMCC 2024.086; NCI-2025-01196 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HUM00254795 (Other: University of Michigan)
Record Dates: First submitted 2025-04-15; First posted 2025-04-23 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Hematopoietic and Lymphatic System Neoplasm; Malignant Solid Neoplasm
MeSH Terms: interventions — Behavior Therapy; Practice Guidelines as Topic; Standard of Care; Health Promotion; Educational Status; Interviews as Topic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Supportive Care (eTAU) (Active Comparator): Patients receive eTAU and receive an educational book to address emotional challenges associated with cancer and strategies and resources to address these challenges over 4-8 weeks on study. Additionally, patients receive check in calls from clinicians QW to answer any questions patients may have about the book.
  Interventions: Other: Best Practice; Other: Communication Intervention; Other: Health Promotion and Education; Other: Questionnaire Administration
- Supportive Care (SFBT-C) (Experimental): Patients undergo virtual SFBT sessions over 30 minutes each QW over 4-8 weeks on study. Patients also receive an educational manual and participate in discussions after each session on study.
  Interventions: Behavioral: Behavioral Intervention; Other: Discussion; Other: Health Promotion and Education; Other: Interview; Other: Questionnaire Administration

INTERVENTIONS:
Behavioral: Behavioral Intervention — Undergo SFBT-C
  Other Names: Behavior Conditioning Therapy; Behavior Modification; Behavior or Life Style Modifications; Behavior Therapy; Behavioral Interventions; Behavioral Modification; Behavioral Therapy; Behavioral Treatment; Behavioral Treatments
  Arms: Supportive Care (SFBT-C)
Other: Best Practice — Receive eTAU
  Other Names: standard of care; standard therapy
  Arms: Supportive Care (eTAU)
Other: Communication Intervention — Receive check in calls from clinician
  Arms: Supportive Care (eTAU)
Other: Discussion — Participate in discussions
  Other Names: Discuss
  Arms: Supportive Care (SFBT-C)
Other: Health Promotion and Education — Receive educational manual
  Arms: Supportive Care (SFBT-C)
Other: Health Promotion and Education — Receive educational book
  Arms: Supportive Care (eTAU)
Other: Interview — Ancillary studies
  Arms: Supportive Care (SFBT-C)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial evaluates the how well a virtually delivered solution-focused brief therapy (SFBT-C) works to decrease adolescent and young adult cancer survivors' psychological distress in comparison to enhanced treatment-as-usual care. Cancer and its treatment can have immediate and long-term impacts on adolescent and young adult cancer survivor's lives, including education and employment, financial stability, sexual health, and social, romantic, and family relationships. Consequently, many adolescent and young adult cancer survivors report psychological distress, often manifesting as depression and anxiety, and may benefit from psychotherapy to improve their engagement with medical treatment and overall quality of life. SFBT-C is a theory-driven and brief hope-based psychotherapy designed for the unique psychosocial needs facing adolescent and young adult cancer survivors. Undergoing SFBT-C may work better than treatment-as-usual care for the support of psychological distress in adolescent and young adult cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* 15 - 39 years old
* Diagnosed with cancer
* Receiving active cancer care (6 weeks post initial diagnosis to control for emotional responses to normative stressors) or within 5 years of post-treatment survivorship
* Experiencing psychological distress (i.e., a t-score >= 57 on the Brief Symptom Inventory - 18 items [BSI-18])
* Fluent in English

Exclusion Criteria:

* End-of-life care
* > 5 years into the post-treatment survivorship
* Major physical challenges (e.g., hearing loss, developmental delay)
* Acute mental health conditions (e.g., active psychosis, suicide risk)
* Receiving or newly initiated psychotherapy for psychological distress during the study period

Ages: 15 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-23 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of solution-focused brief therapy in cancer survivors (SFBT-C) | At baseline, immediate post-intervention, and 4 and 8 weeks post-intervention
  The primary analysis will be a linear regression model with the change score from baseline (T1) to 4 weeks post-intervention completion (T3) in participants' Brief Symptom Inventory, 18-item (BSI-18) t-score as the dependent variable, the intervention assignment, and the randomization strata (age and sex) as the independent variables, i.e., covariates to control for.

SECONDARY OUTCOMES:
Patient's level of hope | Baseline to 8 weeks
  Will be measured using Snyder's Hope Scale (SHS). Will use structural equation modeling (in Mplus) to perform mediation analysis. The primary analysis will be a simple mediation model with the T1 to 8 weeks post-intervention (T4) BSI-18 change score as the dependent variable, treatment assignment as the independent variable, and SHS at immediate post-intervention (T2) as the mediator. An estimated indirect effect (i.e., joint significance testing with bootstrapped standard error) will be computed, and its corresponding 95% confidence interval will determine if hope is a significant treatment mediator.
Quality of life | At baseline, immediate post-intervention, and 4 and 8 weeks post intervention
  Measured by Patient Reported Outcomes Measurement Information System-29 Profile version 2.0. The primary analysis will be a linear regression model with the change score from T1 to T3 (4-week post) in participants' BSI-18 t-score as the dependent variable, the intervention assignment, and the randomization strata (age and sex) as the independent variables, i.e., covariates to control for.

CONTACTS AND LOCATIONS:
Overall Officials: Anao Zhang, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
We will share the study protocol, statistical analysis plan, and analytic codes after a reasonable request and with the discretion of the PI